CLINICAL TRIAL: NCT05714488
Title: Study: A Prospective Evaluation of the Blue Halo BioMedical, LLC "Blue Halo Coil Catheter" for Patients With Prostatic Obstruction
Brief Title: Evaluation of the "Blue Halo Coil Catheter" for Patients With Prostatic Obstruction
Acronym: BlueHaloCoil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blue Halo Biomedical, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-010.3
Record Dates: First submitted 2022-09-20; First posted 2023-02-06 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: The Investigators are conducting a single-arm study with one-group posttest only design.Although this study is a non-randomized control trial, the one-arm design avoids selection and treatment diffusion (among other things). The comparator for the coil catheter is inferior and known to cause injury and infection. Therefore, researchers could not ethically randomly assign subjects to a control group that would receive the alternative device for the sake of comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Blue Halo Coil Catheter for Urinary Retention (Experimental): The indication for use of the Blue Halo Coil Catheter is to facilitate bladder drainage in adult male patients with urinary retention due to benign prostatic hyperplasia. The device is inserted for temporary use up to 28 days.
  Interventions: Device: blue halo coil catheter

INTERVENTIONS:
Device: blue halo coil catheter — device inserted with coil at the bladder and straight arm in the prostatic urethra proximal to the external sphincter

SUMMARY:
The Investigators will study a device for men in urinary retention secondary to Benign Prostatic Hyperplasia, BPH ,who are catheter dependent or who have a Post Void Residual > 350cc. The hypothesis is that the device will allow these participants to return to volitional voiding with a Post Void Residual <75 cc.

DETAILED DESCRIPTION:
The indication for use of the Blue Halo Coil Catheter is to facilitate bladder drainage in adult male patients with urinary retention due to benign prostatic hyperplasia. The device is inserted for temporary use up to 28 days.

Study participants will have a history of Foley catheter use or self-catheterization to drain their bladder.Participants may include men in urinary retention with no prior intervention.

The hypothesis is that the Blue Halo Coil Catheter will reduce the post void residual to <75 cc with volitional voiding.

The Blue Halo Coil Catheter is comprised of a Coiled Retention portion with a guidewire accommodating tip, a short prostate catheter segment, and a pusher/delivery catheter segment, that when left in place allows for the temporary collection of urine prior to conversion to short segment without an external collection device. The tip of the Blue Halo Coil Catheter utilizes a horizontal coil retention device. A monofilament suture is attached to the prostate catheter segment to allow for ease of positioning and removal. The suture also allows for repositioning should the device slip back into the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects > 50 years of age
* Able to provide consent
* Participants in urinary retention with post void residual > 350 cc
* Urinary retention is due to BPH with a prostate volume > 50cc or a prostatic urethral length of 5+ cm
* Subjects with a PSA > 4 ng/ml and a PSA density of 0.1 or less
* Subjects on alpha- blocking drugs or 5-alpha-reductase inhibitor drugs may be included

Exclusion Criteria

* Inability to undergo bladder catheterization ( i.e. urethral stricture)
* Presence of gross hematuria
* Lack of cognitive ability to give consent or keep appointments
* History of Prostate Cancer
* Subject with a PSA > 4 ng/ml and a PSA density of > 0.1 will require prostate biopsy to rule out prostate cancer in order to be considered for study enrollment
* A subject with a prostate nodule will require biopsy to exclude cancer diagnosis
* Subject with a PSA > 10 ng/ml
* Subject taking LHRH analogs or anti-androgen drugs

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — biological males with BPH
Enrollment: 95 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The change in Post Void Residual from baseline to day 28 will be measured and reported | 28 days
  The primary effectiveness endpoint of the study is the number of subjects who were able to return to volitional voiding with a post void residual less then 75 cc during a 28-day study period.Post Void Residual will be measured by bladder ultrasound and reported as cc.

SECONDARY OUTCOMES:
Primary safety endpoint adverse event and device removal | 28 days
  The primary safety endpoint is the number of subjects who had an adverse event related to the Coil Catheter and required removal of the Coil Catheter with an alternative method to drain the bladder, such as an indwelling Foley catheter, or self-intermittent catheterization.
Secondary Safety Endpoint 1, incidence of device encrustation at removal | 28 days
  The number of Blue Halo Coil Catheters that were visibly encrusted at the time of removal
Secondary Safety Endpoint 2,urinary obstruction due to device migration | 28 days
  The number of participants who experienced urinary obstruction secondary to migration of the Blue Halo Coil Catheter, and required replacement of the device
Secondary Safety Endpoint 3, incidence of clinically significant hematuria | 28 days
  The number of participants who experienced clinically significant gross hematuria that necessitated removal of the Blue Halo Coil Catheter and placement of a Foley catheter for bladder drainage

OTHER OUTCOMES:
Bacterial Infection Monitoring | 56 days
  Infection status at the time of insertion and removal of the device will be recorded during the study. Urine culture and sensitivity will be obtained prior to device insertion, at the 28 day removal, and at day 56 follow-up safety visit. The results will be reported as colony forming units, CFU, per ml. Asymptomatic colonization as well as symptomatic Urinary tract infection, UTI, will be reported.
Trends in Renal Function | 56 days
  Serum Creatinine measured as mg/dl will be measured prior to placement of the Blue Halo Coli Catheter, and repeated at the 28 day device removal and at the day 56 follow-up safety visit. This outcome is to observe if there are any changes in renal function that might be attributable to the device
Quality of Life Measurement, no scale to report | 28 days
  The SF-8, Short Form- 8 question survey, will be recorded at the screening visit and the 28 day device removal, to observe any change in Quality of Life issues.
Urinary Bother Inventory, no scale to report | 56 days
  An IRB approved, 4 question, urinary symptom assessment will be recorded at the screening visit, at the 28 day device removal, and at the 56 day safety follow-ip visit.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The University of Alabama-Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Florida Urology Partners, Brandon, Florida
  - Vero Urology Center, Vero Beach, Florida

IPD SHARING:
Plan to Share IPD: Yes
any Adverse Event (AE), Unanticipated AE will be shared with other researchers
Supporting Information: CSR
Time Frame: within 5 days of event and for duration of the study
Access Criteria: all investigators will be emailed by the sponsor with the Adverse Event shared information

REFERENCES:
- [Result] Fontanarosa PB, Roush WR. Acute urinary retention. Emerg Med Clin North Am. 1988 Aug;6(3):419-37. PMID 3292220
- [Result] Samm BJ, Dmochowski RR. Urologic emergencies. Conditions affecting the kidney, ureter, bladder, prostate, and urethra. Postgrad Med. 1996 Oct;100(4):177-80, 183-4. doi: 10.3810/pgm.1996.10.100. PMID 8858090
- [Result] Andersen JT, Nickel JC, Marshall VR, Schulman CC, Boyle P. Finasteride significantly reduces acute urinary retention and need for surgery in patients with symptomatic benign prostatic hyperplasia. Urology. 1997 Jun;49(6):839-45. doi: 10.1016/s0090-4295(97)00185-4. PMID 9187688
- [Result] de la Rosette JJ, Beerlage HP, Debruyne FM. Role of temporary stents in alternative treatment of benign prostatic hyperplasia. J Endourol. 1997 Dec;11(6):467-72. doi: 10.1089/end.1997.11.467. PMID 9440858
- [Result] Williams G. Stents in the lower urinary tract. European Urology Update Series 1992. Vol l (1), p 82-87.
- [Result] Devonec M, Dahlstrand C. Temporary urethral stenting after high-energy transurethral microwave thermotherapy of the prostate. World J Urol. 1998;16(2):120-3. doi: 10.1007/s003450050037. PMID 12073225
- [Result] Feneley RC, Hopley IB, Wells PN. Urinary catheters: history, current status, adverse events and research agenda. J Med Eng Technol. 2015;39(8):459-70. doi: 10.3109/03091902.2015.1085600. Epub 2015 Sep 18. PMID 26383168
- [Result] Hammond, G. A Prospective Evaluation of the Catheter Science M3 "Mini Catheter" for Patients with Prostatic Obstruction. AUA Poster Presentation MP73-06, San Francisco, California, May, 2018
- [Result] Sabharwal S, Sabharwal S. Using Temporary Prostatic Stents to Eliminate Bacterial Colonization in Men with Chronic Indwelling Catheters: A Pilot Study. Cureus. 2018 Aug 16;10(8):e3152. doi: 10.7759/cureus.3152. PMID 30410822
- [Result] Garcia MM, Gulati S, Liepmann D, Stackhouse GB, Greene K, Stoller ML. Traditional Foley drainage systems--do they drain the bladder? J Urol. 2007 Jan;177(1):203-7; discussion 207. doi: 10.1016/j.juro.2006.08.101. PMID 17162043
- [Result] Shore ND, Dineen MK, Saslawsky MJ, Lumerman JH, Corica AP. A temporary intraurethral prostatic stent relieves prostatic obstruction following transurethral microwave thermotherapy. J Urol. 2007 Mar;177(3):1040-6. doi: 10.1016/j.juro.2006.10.059. PMID 17296408